CLINICAL TRIAL: NCT04742088
Title: Assessment of the Safety and Performance of a Compression Ankle Support in the Prevention of Injuries During Sports Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ankleSOFT100
Record Dates: First submitted 2020-09-04; First posted 2021-02-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain; Chronic Instability of Ankle Joint
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthosis group (Experimental)
  Interventions: Device: ankleSOFT100

INTERVENTIONS:
Device: ankleSOFT100 — During the first two weeks of follow-up, the subject shall not use the device during the sports sessions. The subject shall use the device during the sports sessions for the next 4 weeks (6 weeks of follow-up)

SUMMARY:
Decathlon has developed ankleSOFT100 product which is medical device designed to reduce pain and joint instability during sport practice. The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon ankleSOFT100 product to demonstrate safety and performance of this device in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥18 years old
* Subject has chronic pain AND / OR chronic ankle instability
* The current condition of his/her ankle allows the subject to pursue a usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (6 weeks)
* Subject is affiliated to the French social security regime

Non-inclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (ankle brace or articulated orthosis) during sports sessions during the last month
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, elastodiene, elastane, polyester, synthetic rubber)
* Adult subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Functional score | At baseline and 6 weeks of follow-up
  Change from baseline functional result (Cumberland Ankle Instability Tool: 0-30 points) at 6 weeks

SECONDARY OUTCOMES:
Confidence level | At baseline and 6 weeks of follow-up
  Gap in the confidence level (patient rated outcome with 6 questions, ranging from 0 to 100) related to physical activity, between the baseline and last follow-up visit
Ankle instability | At 2 weeks and 6 weeks of follow-up
  Comparison of ankle instability between the first two weeks of follow-up (without use of the device during sports sessions) and the following four weeks (with use of the device during sports sessions), measured through a Numerical Rating Scale (NRS, ranging from 0 to 10)
Ankle pain | At 2 weeks and 6 weeks of follow-up
  Comparison of ankle pain between the first two weeks of follow-up (without use of the device during sports sessions) and the following four weeks (with use of the device during sports sessions), measured through a NRS (ranging from 0 to 10)
Safety (adverse events) | 6 weeks of follow-up
  Rate of adverse events occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (4):
- France (4):
  - Centre de rééducation et de balnéothérapie Kinés Faches, Faches-Thumesnil
  - Centre Hospitalier Universitaire de Lille, Lille
  - Cabinet de kinésithérapie du Belvédère, Paris
  - KOSS Paris 8, Paris

IPD SHARING:
Plan to Share IPD: No